CLINICAL TRIAL: NCT05720507
Title: Cafe Move: A Novel Program for Prevention of Age-Related Physical Frailty
Brief Title: Preliminary Testing of Cafe Move for Primary Prevention of Physical Frailty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 76-22
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Aging
Keywords: Frailty; Physical function; Strength; Mobility; Balance
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Single cohort double baseline design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Cafe Move — Participants will be offered the opportunity to choose from a number of physical function assessments and subsequently provided personalized reports of performance results.

SUMMARY:
This project explores a novel means of health promotion and prevention of age-related physical frailty, which is designed to overcome barriers to access and promote autonomy in managing physical health.

DETAILED DESCRIPTION:
The purpose of this investigation is to field-test a physical function assessment paradigm, designed to inform people of their physical function relative to peers of similar demographic characteristics (e.g., similar age, sex, height, etc.), to promote recommended preventive health behaviors. The physical function assessment paradigm is known as Cafe Move. Our primary research hypothesis is that people will advance along the stages of behavior change (i.e., more likely to participate in recommended preventive healthcare for physical function), after accessing Cafe Move assessments. This study is a single cohort (n=36 participants), double-baseline design, intended primarily to collect pilot data. The results will inform the design of a larger controlled trial.

This study will examine the safety, feasibility, acceptability, and preliminary efficacy of Café Move. Briefly, we will make Café Move available to at-risk populations (i.e., independent-living older adults) via the following approach. First, during a 3-month control phase, we will monitor participants' health behaviors and engagement with preventive health offerings via periodic phone surveys. We will then make Café Move available and subsequently monitor health behaviors and engagement with preventive health offerings. This design will allow us to examine feasibility of the Café Move intervention, to better understand the reach of the program within and across communities, and to determine variance and covariance for the outcome measures of interest.

ELIGIBILITY:
Inclusion Criteria:

* Legally autonomous to consent
* Lives independently
* Ability to sit, stand, and walk without the assistance of another person

Exclusion Criteria:

* Not legally autonomous to consent
* Institutionalized

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Health Behavior Stages of Change Questionnaire | through study completion, average of 4-6 months
  Self-reported measure of engagement with preventive care or wellness activities

SECONDARY OUTCOMES:
Healthcare Access and Utilization Questionnaire | through study completion, average of 4-6 months
  Self-reported measure of healthcare utilization of a number of different services

OTHER OUTCOMES:
Two-minute walk test (2MWT) | through study completion, average of 4-6 months
  Measure of distance walked in 2 minutes along a 50-foot course
Grip Strength | through study completion, average of 4-6 months
  Measure of participants' maximum grip strength using a handheld dynamometer
Postural Sway | through study completion, average of 4-6 months
  Timed test of participants' ability to balance under 4 different conditions
Activities-Specific Balance Confidence Scale | through study completion, average of 4-6 months
  Self-reported questionnaire that assess participants' perceived balance
Lifespace Mobility Questionnaire | through study completion, average of 4-6 months
  Self-reported questionnaire that assess participants' interaction with home and community settings
Role Participation Questionnaire | through study completion, average of 4-6 months
  Self-reported questionnaire that captures various social, demographic, and activity level information from participants
Physical Function Questionnaire | through study completion, average of 4-6 months
  Self-reported questionnaire assessing perceived function with daily activities

CONTACTS AND LOCATIONS:
Locations (1):
- University of Montana, Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: No